CLINICAL TRIAL: NCT05695599
Title: Supervised Whole Body Vibration Training for the Improvement of Body Composition, Microbiota and Physical Fitness After Bariatric Surgery
Brief Title: Whole Body Vibration After Bariatric Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Centro de Investigación Biomédica en Red de Enfermedades Hepáticas y Digestivas (CIBEREHD) (Unknown); Centro de Investigación Biomédica en Red Fisiopatología de la Obesidad y Nutrición (CIBEROBN) (Unknown)
Responsible Party: Principal Investigator, José A. Casajús, Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBVBS
Record Dates: First submitted 2022-12-19; First posted 2023-01-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Bariatric Surgery and Whole Body Vibration Training; Bariatric Surgery
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will only have codes but in the database but will not know which code corresponds to which group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration (Experimental): Participants will undergo a whole body vibration training
  Interventions: Device: Whole body vibration training
- Control Group (No Intervention): Participants will not perform an intervention

INTERVENTIONS:
Device: Whole body vibration training — 3 times per week of 20 to 30 minute sessions during 16 weeks of training
  Other Names: Exercise
  Arms: Whole body vibration

SUMMARY:
Morbid obesity is defined as a complex chronic condition in which a person presents a body mass index above 40 kg/m2. This disease increases the risk of several co-morbidities and entails a reduction in life expectancy of 10 years. Its prevalence is increasing in developed countries and bariatric surgery has been suggested to be one of the best tools to counteract it. Nonetheless, this surgery also presents negative effects such as loss of bone mineral density (BMD) and muscle mass and an increased fracture risk. The aim of the present study is to elucidate the effects of surgery and a whole body vibration training (WBV) on body composition, physical fitness, microbiota and cardiometabolic markers. Twenty eight participants will undergo bariatric surgery and will be randomly allocated into a control group or a WBV group. The whole body vibration group will have a duration of 4 months in which participants will train three times per week (30 minutes per session). Measurements of body composition (dual energy x-ray and peripheral quantitative computed tomography), physical fitness (muscular strength, aerobic fitness and balance), gait biomechanics, cardiometabolic markers, gut microbiota, quality of life and physical activity levels will be registered in four different timepoints (1. Before the intervention, 2) 45 days after the surgery, 3) Six months after the surgery, and 4) 18 months after the surgery. The cost of the surgery and the exercise program will also be calculated to perform a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are going to undergo Roux-en-Y gastric bypass with a Body mass index above 40 and below 180 kg.
* With an age between 18 and 50 years of age
* Living in the city of Zaragoza

Exclusion Criteria:

* History of cancer in the last 5 years
* Have a pacemaker or being diagnosed with a cardiac problem that disables the participant to take place in an exercise program
* To have suffered an acute myocardial infarction in the last 6 months
* To present uncontrolled hypertension
* Fracture in the last year
* Any other condition that the physician deems as a contraindication for performing supervised physical exercise
* Menopause

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | pre-surgery
  Bone density measured with dual energy x-ray
Bone mineral density | 2 months post-surgery
  Bone density measured with dual energy x-ray
Bone mineral density | 6 months post-surgery
  Bone density measured with dual energy x-ray
Bone mineral density | 18 months post-surgery
  Bone density measured with dual energy x-ray
Bone structure | pre-surgery
  Radius strength and structure measured with peripheral quantitative computed tomography
Bone structure | 2 months post-surgery
  Radius strength and structure measured with peripheral quantitative computed tomography
Bone structure | 6 months post-surgery
  Radius strength and structure measured with peripheral quantitative computed tomography
Bone structure | 18 months post-surgery
  Radius strength and structure measured with peripheral quantitative computed tomography
Body composition | pre-surgery
  Body fat and visceral adipose tissue measured with Dual energy X-ray
Body composition | 2 months post-surgery
  Body fat and visceral adipose tissue measured with Dual energy X-ray
Body composition | 6 months post-surgery
  Body fat and visceral adipose tissue measured with Dual energy X-ray
Body composition | 18 months post-surgery
  Body fat and visceral adipose tissue measured with Dual energy X-ray
Fecal gut microbiota | pre-surgery
  Stool specimens will be taken. Samples will be sequenced by Shallow Shotgun Metagenomic sequencing using Illumina Sequencing PE150 (5 G raw data per sample).
Fecal gut microbiota | 6 months post-surgery
  Stool specimens will be taken. Samples will be sequenced by Shallow Shotgun Metagenomic sequencing using Illumina Sequencing PE150 (5 G raw data per sample).
Fecal gut microbiota | 18 months post-surgery
  Stool specimens will be taken. Samples will be sequenced by Shallow Shotgun Metagenomic sequencing using Illumina Sequencing PE150 (5 G raw data per sample).

SECONDARY OUTCOMES:
Basal metabolic rate | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Basal metabolic rate
Heart rate variability | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Heart rate variability measured in fasting and resting conditions
Aerobic capacity | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Bruce protocol on a treadmill
Muscular strength of the upper limbs | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Measured with a handgrip dynamometer
Muscular strength of the lower limbs | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Measured with the stand and sit chair test
Agility | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Measured with the time up and go test. Sitting on a chair the participant has to stand up and walk 2,4 meters forward, turn and sit back on the chair.
Balance | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Measured with the SPPB battery in three different position (feet together, tandem, semi tandem)
Gait kinematics | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Gait kinematics measured with inertial sensors
Frailty status | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  SPPB measures
Quality of life of participants SF36 | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Quality of life measured with the SF36
Quality of life of participants EUROQOL 5Q | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Quality of life measured with the EUROQOL 5Q
Pain scale | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Pain measured with the WOMAC questionnaire
Objective physical activity levels | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Physical activity levels registered with triaxial accelerometers that they will wear during 7 days.
Physical activity levels | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Physical activity levels measures with IPAQ-short
Ankle range of motion | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Measurement of dorsiflexion and plantar flexion
Inflammatory markers | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Interleukin 6, TNF alpha, and reactive C protein
Blood glucose | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Glucose levels
Cholesterol | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Blood cholesterol levels (LDL and HDL)
Insulin resistance | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  HOMA test and insulin levels
Kidney markers | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Creatinine levels
Liver function (ALT) | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Alanine transaminase levels
Liver function (AST) | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Aspartate transaminase
Liver function (ALP) | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Alkaline phosphatase
Liver function (GGT) | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Gamma-glutamyl transferase
Liver function (bilirubin) | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Serum bilirubin levels
International normalised ratio test | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  INR coagulation
Albumin levels | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Serum albumin levels
Iron metabolism | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Iron metabolism markers
Vitamin B12 levels | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Plasma vitamin B12 levels
Folic acid levels | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Plasma folic acid levels
Hydroxyvitamin D | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Plasma Hydroxyvitamin D levels
Calcium | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Plasma calcium levels
Phosphorus | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Plasma phosphorus levels
Parathyroid hormone | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Parathyroid hormone plasma levels
Bone alkaline phosphatase | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Bone alkaline phosphatase plasma levels
Leptin | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Leptin plasma levels
Adinopectin | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Adinopectin plasma levels
Diet | pre-surgery, 6 months post-surgery
  Diet will be assessed though a food frequency questionnaire
Depression, anxiety and stress questionnaire | pre-surgery, 2 months post-surgery, 6 months post-surgery and 18 months post-surgery
  Dass 21 scale

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - GENUD Research group, Zaragoza
  - Hospital Clinic Universitario, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Bruton A, Irun P, Matute-Llorente A, Lozano-Berges G, Moradell A, Ara-Gimeno S, Subias-Perie J, Sanchez-Luengo M, Hijos-Mallada G, Garcia-Mateo S, Arechavaleta S, Palacios Fanlo MJ, Lanas A, Casajus JA. Effects of whole-body vibration on body composition, microbiota, cardiometabolic markers, physical fitness, and quality of life after bariatric surgery: protocol for a randomized controlled trial. Trials. 2024 Jun 26;25(1):413. doi: 10.1186/s13063-024-08221-7. PMID 38926901